CLINICAL TRIAL: NCT01686100
Title: CT-angiographic Follow Upp of Patients That Underwent Coronary Bypass Surgery Between 1993-1997. A Randomized Longitudinal Trial.
Brief Title: CT-angiographic Follow up of Patients That Underwent Coronary Bypass Surgery Between 1993-1997
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro County Council (Other Government)
Responsible Party: Principal Investigator, Ninos Samano M.D., Doctor, Örebro County Council
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 102841
Record Dates: First submitted 2012-09-12; First posted 2012-09-17 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery bypass grafting; Saphenous vein grafts
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- No touch vein grafts (Active Comparator): The grafts were harvested with there surrounding tissues.
  Interventions: Procedure: No touch technique
- Conventional vein grafts. (Active Comparator): The grafts were stripped from surrounding tissue.
  Interventions: Procedure: Conventional technique

INTERVENTIONS:
Procedure: No touch technique — The vein graft is harvested with its surronding tissues.
  Arms: No touch vein grafts
Procedure: Conventional technique — The vein graft is stripped from its surrounding tissues.
  Arms: Conventional vein grafts.

SUMMARY:
Coronary artery surgery (CABG) is necessary to improve blood circulation in many patients with coronary artery disease. This is done by using alternative blood vessels (grafts) to bypass the stenosed coronary arteries. In CABG, vein grafts are traditionally used where surrounding tissue is removed, this may damage the vessel and influence its patency.

The "no-touch" technique was developed by Professor Domingos Souza at the Department of Cardiovascular and Thoracic Surgery, Örebro University Hospital. This technique includes taking out the vein with its surrounding tissue and by this way the vessel is less damaged. The first two follow ups have shown that no-touch grafts had better patency than conventionally extracted graft at 18 months and 8.5 years.

This long term follow up is a continuation of the randomized trial started in 1993 where the patency and incidence of stenoses in the no touch and conventional vein grafts has been studied.

ELIGIBILITY:
Inclusion Criteria:

1. First time coronary artery bypass grafting with either conventional or no touch vein grafts performed by Dr.Souza between 1993-1997.
2. Included in the previous follow up studies
3. Signed and dated consent.

Exclusion Criteria:

1. Allergy to contrast
2. Renal failure
3. Uncontrolled diabetes
4. Unable to implement the study according to protocol -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Patency of the grafts | Mean time of 15 years.

SECONDARY OUTCOMES:
Stenosis in the grafts. | Mean time of 15 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Cardiovascular and Thoracic Surgery, Örebro University Hospital, Örebro, Sweden

REFERENCES:
- [Background] Souza DS, Johansson B, Bojo L, Karlsson R, Geijer H, Filbey D, Bodin L, Arbeus M, Dashwood MR. Harvesting the saphenous vein with surrounding tissue for CABG provides long-term graft patency comparable to the left internal thoracic artery: results of a randomized longitudinal trial. J Thorac Cardiovasc Surg. 2006 Aug;132(2):373-8. doi: 10.1016/j.jtcvs.2006.04.002. PMID 16872965
- [Background] Loesch A, Dashwood MR, Souza DS. Does the method of harvesting the saphenous vein for coronary artery bypass surgery affect venous smooth muscle cells? iNOS immunolabelling and ultrastructural findings. Int J Surg. 2006;4(1):20-9. doi: 10.1016/j.ijsu.2005.11.002. Epub 2006 Jan 3. PMID 17462310
- [Background] Dashwood MR, Dooley A, Shi-Wen X, Abraham DJ, Dreifaldt M, Souza DS. Perivascular fat-derived leptin: a potential role in improved vein graft performance in coronary artery bypass surgery. Interact Cardiovasc Thorac Surg. 2011 Feb;12(2):170-3. doi: 10.1510/icvts.2010.247874. Epub 2010 Nov 3. PMID 21051379
- [Background] Dreifaldt M, Souza DS, Loesch A, Muddle JR, Karlsson MG, Filbey D, Bodin L, Norgren L, Dashwood MR. The "no-touch" harvesting technique for vein grafts in coronary artery bypass surgery preserves an intact vasa vasorum. J Thorac Cardiovasc Surg. 2011 Jan;141(1):145-50. doi: 10.1016/j.jtcvs.2010.02.005. Epub 2010 Apr 9. PMID 20381817
- [Background] Johansson BL, Souza DS, Bodin L, Filbey D, Loesch A, Geijer H, Bojo L. Slower progression of atherosclerosis in vein grafts harvested with 'no touch' technique compared with conventional harvesting technique in coronary artery bypass grafting: an angiographic and intravascular ultrasound study. Eur J Cardiothorac Surg. 2010 Oct;38(4):414-9. doi: 10.1016/j.ejcts.2010.02.007. Epub 2010 Apr 1. PMID 20362457
- [Background] Johansson BL, Souza DS, Bodin L, Filbey D, Bojo L. No touch vein harvesting technique for CABG improves the long-term clinical outcome. Scand Cardiovasc J. 2009 Feb;43(1):63-8. doi: 10.1080/14017430802140104. PMID 18609044
- [Background] Rueda Fd, Souza D, Lima Rde C, Menezes A, Johansson B, Dashwood M, The E, Gesteira M, Escobar M, Vasconcelos F. Novel no-touch technique of harvesting the saphenous vein for coronary artery bypass grafting. Arq Bras Cardiol. 2008 Jun;90(6):356-62. doi: 10.1590/s0066-782x2008000600002. English, Portuguese. PMID 18592087
- [Background] Dashwood MR, Savage K, Dooley A, Shi-Wen X, Abraham DJ, Souza DS. Effect of vein graft harvesting on endothelial nitric oxide synthase and nitric oxide production. Ann Thorac Surg. 2005 Sep;80(3):939-44. doi: 10.1016/j.athoracsur.2005.03.042. PMID 16122459
- [Background] Dashwood M, Anand R, Loesch A, Souza D. Surgical trauma and vein graft failure: further evidence for a role of ET-1 in graft occlusion. J Cardiovasc Pharmacol. 2004 Nov;44 Suppl 1:S16-9. doi: 10.1097/01.fjc.0000166222.50346.c6. PMID 15838269
- [Background] Souza DS, Dashwood MR, Tsui JC, Filbey D, Bodin L, Johansson B, Borowiec J. Improved patency in vein grafts harvested with surrounding tissue: results of a randomized study using three harvesting techniques. Ann Thorac Surg. 2002 Apr;73(4):1189-95. doi: 10.1016/s0003-4975(02)03425-2. PMID 11996262
- [Background] Tsui JC, Souza DS, Filbey D, Karlsson MG, Dashwood MR. Localization of nitric oxide synthase in saphenous vein grafts harvested with a novel "no-touch" technique: potential role of nitric oxide contribution to improved early graft patency rates. J Vasc Surg. 2002 Feb;35(2):356-62. doi: 10.1067/mva.2002.121072. PMID 11854735
- [Background] Tsui JC, Souza DS, Filbey D, Bomfim V, Dashwood MR. Preserved endothelial integrity and nitric oxide synthase in saphenous vein grafts harvested by a 'no-touch' technique. Br J Surg. 2001 Sep;88(9):1209-15. doi: 10.1046/j.0007-1323.2001.01855.x. PMID 11531869
- [Background] Souza DS, Christofferson RH, Bomfim V, Filbey D. "No-touch" technique using saphenous vein harvested with its surrounding tissue for coronary artery bypass grafting maintains an intact endothelium. Scand Cardiovasc J. 1999;33(6):323-9. doi: 10.1080/14017439950141362. PMID 10622542
- [Background] Souza D. A new no-touch preparation technique. Technical notes. Scand J Thorac Cardiovasc Surg. 1996;30(1):41-4. doi: 10.3109/14017439609107239. No abstract available. PMID 8727856
- [Derived] Samano N, Geijer H, Liden M, Fremes S, Bodin L, Souza D. The no-touch saphenous vein for coronary artery bypass grafting maintains a patency, after 16 years, comparable to the left internal thoracic artery: A randomized trial. J Thorac Cardiovasc Surg. 2015 Oct;150(4):880-8. doi: 10.1016/j.jtcvs.2015.07.027. Epub 2015 Jul 15. PMID 26282605
- [Derived] Johansson B, Samano N, Souza D, Bodin L, Filbey D, Mannion JD, Bojo L. The no-touch vein graft for coronary artery bypass surgery preserves the left ventricular ejection fraction at 16 years postoperatively: long-term data from a longitudinal randomised trial. Open Heart. 2015 Mar 24;2(1):e000204. doi: 10.1136/openhrt-2014-000204. eCollection 2015. PMID 25852948